CLINICAL TRIAL: NCT07098169
Title: Randomized Clinical Trial of iTEST: A Blended Intervention Targeting Introspective Accuracy
Acronym: iTEST R33
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); The University of Texas at Dallas (Other); University of Miami (Other)
Responsible Party: Principal Investigator, Colin Depp, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4R33MH129379 (NIH)
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia Disorders; Schizoaffective Disorder; Psychotic Disorder
Keywords: Digital health; Cognitive training; Schizophrenia; Psychosis; Functional rehabilitation
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: Parallel arm randomized
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iTEST (Experimental): iTEST includes 6 weeks of weekly coaching sessions that last for 60 minutes each delivered by telehealth or in person per the participant's preference, followed by 3 bi-weekly 30 minute booster telephone calls. ITEST also includes daily cognitive tasks that involve task of memory for words or recognizing facial emotions. Participants guess the number correct after each task and are provided feedback on the accuracy of their guesses. These tasks occur once per day days per week and continue occur over 12 weeks.
  Interventions: Behavioral: iTEST
- Active Control (Active Comparator): The control condition includes 6 weeks of weekly coaching sessions that last for 60 minutes each delivered by telehealth or in person per the participant's preference, followed by 3 bi-weekly 30 minute booster telephone calls. Participants also complete daily cognitive tasks that involve task of memory for words or recognizing facial emotions. Participants are provided feedback their performance. These tasks occur once per day days per week and continue occur over 12 weeks.
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: iTEST — iTEST is a computerized training intervention delivered on a mobile device that is coupled with individual contacts with a therapist/coach. The mobile components train in improving participant's ability to form accurate judgments about their performance and their rate of functional activities. The intervention involves coaching coupled with automated training that is delivered on a mobile device. The automated training involves daily cognitive tests in which the goal for treatment is to improve judgments of accuracy of self-assessment, and coaching is aimed at applying improving metacognitive awareness to every day activities. i
  Arms: iTEST
Behavioral: Active Control — Behavioral: Mobile cognitive tests will be administered to control subjects. Participants will receive feedback regarding their performance but not on the accuracy of their self-ratings. Coaching will also be coupled with mobile cognitive tests and will include goal-setting without specific mention of Introspective Accuracy (IA). in place of content related to IA, participants will receive psychoeducation about the benefits of sleep, physical activity, and social connection to overall cognitive health
  Arms: Active Control

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a psychosocial intervention called iTEST for people with psychotic disorders that targets introspective accuracy, or the ability to accurately gauge ones abilities. iTEST combines daily cognitive training on a mobile device with coaching that addresses recovery goals. In this trial, we will randomize people to one of two interventions conditions, iTEST or a control condition that receives coaching and cognitive training that does not emphasize introspective accuracy. Both interventions will take place over 12 weeks and participants will be asked to complete assessments at baseline, 6 weeks, 12 weeks, and 24 weeks. The primary outcome of the study is community functioning. Participants will be from three metropolitan areas: San Diego, Dallas, or Miami.

DETAILED DESCRIPTION:
This NIH-supported clinical trial is the second phase of a two-phase program, funded by Development of Psychosocial Therapeutic and Preventive Interventions for Mental Disorders, R61/R33. The overarching goal of this second R33 phase is to evaluate the replicability of R61 findings in a larger randomized control trial with iTEST, a new blended mobile intervention that is aimed at improving introspective accuracy (IA) in people with psychotic disorders, vs. a control condition that is time-equivalent but does not train in introspective accuracy. Introspective accuracy is the degree to which one's self-assessment of performance or abilities corresponds with objective data. Recent research indicates that poor IA is an independent predictor of functional disability. Yet, there are currently no treatments that directly target IA. Basic experimental research and other lines of evidence suggest IA is malleable, and that improvement in task-based IA transfers to untrained tasks. The investigators have developed and completed usability testing of iTEST, a novel blended IA targeted mobile intervention. iTEST integrates graduated drill-and-practice training in IA delivered on a mobile device with personalized coaching in applying IA to everyday compensatory behaviors. In the R61 open trial phase, people with psychotic disorders with at least minimal functional impairment were recruited and found that the intervention led to clinically significant changes in task-based IA along with transfer to an untrained task (target mechanisms). It was determined that the dose of intervention needed to achieve clinically significant improvement in IA targets was achieved at 12 weeks. Therefore, in this trial phase R33, the intervention will last for 12 weeks with a 3-month follow-up. A total of 201 persons who are diagnosed with schizophrenia or schizoaffective disorder will be recruited into this trial

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary informed consent to participate and capacity to consent as measured by the UCSD Brief Assessment of Capacity to Consent (UBACC)
2. Age 18 to 65;
3. DSM-5 diagnosis of schizophrenia or schizoaffective disorder based on a structured diagnostic interview and available medical record review;
4. ≥ 6th grade reading level on the Wide Range Achievement Test-4 Reading subtest (needed to read instructions on device);
5. Stable co-treatments (no hospitalizations or medication class changes in 2 months before enrollment). The investigators will determine symptom and medication stability by best-estimate history with information from medical records;
6. Availability of a clinician (staff member, case manager, other mental health clinician) or close associate (family member, friend) with at least monthly contact who can be their informant
7. Minimum level of functional impairment based on milestones, excluding participants who are full-time employed and financially responsible for their household.

Exclusion Criteria:

1. Greater than moderate disorganization on the Positive and Negative Syndrome Scale (P2-Disorganization item >5)
2. DSM-5 alcohol or substance dependence in past 3 months based on interview
3. Level of care required interferes with outpatient therapy (e.g., hospitalized; severe medical illness); 4) Unable to adequately see or manually manipulate a smartphone.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Informant-Rated Specific Level of Function (SLOF) Scale | Change from baseline to 3 month follow up
  Measure of participant's community functioning rated by an informant. Scale scores range from 43 to 215 with higher scores reflecting better functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Pinkham, PhD, Principal Investigator — The University of Texas at Dallas
Locations (3):
- United States (3):
  - UC San Diego, San Diego, California
  - University of Miami, Miami, Florida
  - University of Texas at Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from measures administered
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data availability is at the end of the study (2028) and there is no end date
Access Criteria: Qualified researchers who are eligible to access the NDA system

REFERENCES:
- [Result] Berretta SA, Abaya N, Parrish E, McBride LE, Moore RC, Ackerman R, Harvey PD, Pinkham AE, Depp CA. Protocol for evaluation of iTEST, a novel blended intervention to enhance introspective accuracy in psychotic disorders. NPP Digit Psychiatry Neurosci. 2025;3(1):5. doi: 10.1038/s44277-024-00024-7. Epub 2025 Feb 14. PMID 39959603